CLINICAL TRIAL: NCT04234841
Title: Can Thrombosis and Fibrinolysis Markers in Patients Undergoing Aortic Valve Replacement Predict Outcome
Brief Title: Avr Thrombosis OutcoMe Study
Acronym: ATOM
Status: Not yet recruiting | Type: Observational
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RD2019-11
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Aortic Stenosis
Keywords: TAVI; SAVR
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples obtained through phlebotomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Surgical Aortic Valve Replacement (SAVR): This cohort includes patients who will be undergoing surgical aortic valve replacement
  Interventions: Diagnostic Test: Blood test
- Transcatheter Aortic Valve Implantation (TAVI): This cohort includes patients who will be undergoing Transcatheter Aortic Valve Implantation
  Interventions: Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Blood test — Blood test

SUMMARY:
This study aims to utilise novel biomarkers assessing thrombosis and thrombolysis (through a blood test), to identify patients undergoing either surgical aortic valve replacement (SAVR) or transcatheter aortic valve implantation (TAVI) who are at risk of thrombosis, and relate this to clinical thrombotic and thromboembolic adverse events and subclinical valve thrombosis, and identify the timeframe of greatest risk for valve thrombosis.

DETAILED DESCRIPTION:
Recent studies have highlighted the risk of peri-operative thrombosis in patients undergoing aortic valve replacement (AVR) and the subsequent risk of subclinical valve thrombosis in bioprosthetic AVR. The risk is significantly greater with transcatheter aortic valve implantation (TAVI) than surgical aortic valve replacement (SAVR), and can lead to stroke and other neurological events including death, and early valve failure secondary to restricted leaflet mobility.

Whilst oral anticoagulation (OAC) can reduce thrombosis, OAC has been shown to significantly and unacceptably increase the risk of bleeding when applied to all-comers undergoing TAVI. It would therefore be desirable to identify which patients are at increased thrombosis risk so these can be targeted with antithrombotic medications, whilst avoiding unnecessary bleeding risk in low risk patients.

In this study, we will aim to identify those patients at greatest risk of thrombosis using novel biomarkers (assessing thrombosis and thrombolysis), and note whether these tests are able to predict adverse events.

The tests for thrombosis and thrombolysis will involve a blood draw, which will be taken at various time points in the study to signal the time point of greatest thrombogenicity, which may be dependent on anti-platelet and anticoagulant therapy that the patient is prescribed.

Adverse events include MACCE (myocardial infarction, stroke, TIA (transient ischaemic attack) and death), systemic embolism, clinical and subclinical valve thrombosis, valve restriction and bleeding.

4D CT, echocardiography and clinical reviews will be performed at regular time points in the study to identify adverse events. The follow-up for each patent will be 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 years or over.
2. Patients diagnosed with aortic valve disease, undergoing surgical or transcatheter AVR and free of exclusion criteria below.
3. The patient is willing and able to understand the Patient Information Sheet and provide informed consent.
4. The patient agrees to comply with the study protocol, including phlebotomy and imaging as required at pre-specified time points.

Exclusion Criteria:

1. Inability to provide valid informed consent.
2. Male and female patients aged < 18 years of age.
3. The patient has, in the opinion of the investigator, significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, haemorrhagic, metabolic or other disease likely to confound the study requirements or analyses.
4. The patient has a history of substance abuse or demonstrates signs or clinical features of active substance abuse or active psychiatric disease that may result in non-compliance with visits or inability to obtain venous access.
5. Alcohol consumption above recommended safe levels (i.e. more than 14 units per week owing to the potential effects of high alcohol levels on platelet reactivity).
6. Any illness deemed significant by the investigator during the four (4) weeks preceding the screening period of the study such as sepsis.
7. Any major bleeding diathesis or blood dyscrasia (platelets < 70 x 109/l, Hb < 8 g/dl, INR > 1.4, APTT > x 2 UNL, leucocyte count < 3.5 x 109/l, neutrophil count < 1 x 109/l).
8. Currently enrolled in an investigational device or drug trial.
9. Active or disseminated malignancy at the time of recruitment.

   Additionally, for those patients taking part in the additional 4D CT angiography substudy:
10. Any contraindications to CT angiography: renal failure (Cr>250 μmol/L or eGFR<30 mL/min) due to the additional risk of contrast medium nephrotoxicity; or allergy to iodine.
11. Women of childbearing age who have not had a hysterectomy and/or who may be breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing surgical bioprosthetic aortic valve replacement and transcatheter aortic valve implantation
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
MACCE | 5 years (total duration of study)
  Myocardial infarction, Stroke, Transient Ischaemic Attack (TIA), death
Bleeding | 5 years (total duration of study)
  BARC
Systemic embolism | 5 years (total duration of study)

SECONDARY OUTCOMES:
Subclinical valve thrombosis | 5 years (total duration of study)
New/worsening AF | 5 years (total duration of study)

CONTACTS AND LOCATIONS:
Locations (1):
- East and North Hertfordshire NHS Trust, Stevenage, Hertforshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No